CLINICAL TRIAL: NCT00624819
Title: Long-term Follow-up Study to Assess Antibody Persistence in Children Previously Vaccinated With Four Doses of Pneumococcal Conjugate Vaccine in Primary Vaccination Study (105553) and Booster Vaccination Study (107046)
Brief Title: Assessment of Antibody Persistence in Children Previously Vaccinated With Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111345 (Mth 12); 111346 (Mth 24) (Other: GSK); 111347 (Mth 48) (Other: GSK); 2007-005392-34 (EudraCT Number)
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
Keywords: Streptococcus pneumoniae; Haemophilus influenzae; Pneumococcal conjugate vaccine; Antibody persistence
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — PHiD-CV vaccine; Heptavalent Pneumococcal Conjugate Vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Hepatitis A Vaccines

ARMS (4):
- Synflorix + Infanrix + Havrix and/or Varilrix Group (Experimental): This group consisted of subjects primed with Synflorix vaccine in the 10PN-PD-DIT-001 (1105553) and 007 (107046) studies. In 105553 study, subjects had been primed with 3 doses of Synflorix vaccine at 2, 3 and 4 months of age co-administered with Infanrix related vaccines. In 107046 study, subjects had received a booster dose of Synflorix vaccine at 12-18 months of age co-administered with Infanrix hexa vaccine. In this study, in the Year 4 (111347 study), subjects received at Month 48 (4 years post Dose 1 in study 105553) one additional dose of Synflorix vaccine. In addition, subjects were also offered vaccination against hepatitis A (2 doses of Havrix) and/or against varicella (a single dose of Varilrix).
  Interventions: Biological: GSK1024805A; Biological: Infanrix hexa; Biological: Havrix; Biological: Varilrix
- Prevenar + Infanrix + Havrix and/or Varilrix Group (Active Comparator): This group consisted of subjects vaccinated with Prevenar vaccine in the 10PN-PD-DIT-001 (105553) and 007 (107046) studies. In 105553 study, subjects had been primed with 3 doses of Prevenar vaccine at 2, 3 and 4 months of age co-administered with Infanrix related vaccines. In 107046 study, subjects had received a booster dose at 12-18 months of age of Prevenar vaccine co-administered with Infanrix hexa vaccine. In this study, in the Year 4 111347 study, subjects had received at Month 48 (4 years post Dose 1 in study 105553) one dose of Synflorix vaccine. In addition, subjects were also offered vaccination against hepatitis A (2 doses of Havrix and/or against varicella (a single dose of Varilrix).
  Interventions: Biological: Prevenar; Biological: Infanrix hexa; Biological: Havrix; Biological: Varilrix
- Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix (Experimental): This group consisted of subjects vaccinated with Prevenar and Synflorix vaccines in the 10PN-PD-DIT-001 (105553) and 10PN-PD-DIT-007 (107046) studies. In 105553 study, subjects had been primed with 3 doses Prevenar vaccine at 2, 3 and 4 months of age co-administered with Infanrix related vaccines. In the 107046 study, subjects had received at 12-18 months of age a booster dose of Synflorix vaccine co-administered with Infanrix hexa vaccine. In this study, in the Year 4 (111347 study), subjects had received at Month 48 (4 years post Dose 1 in study 105553) one additional dose of Synflorix vaccine. In addition, subjects were also offered vaccination against hepatitis A (2 doses of Havrix and/or against varicella (a single dose of Varilrix).
  Interventions: Biological: GSK1024805A; Biological: Prevenar; Biological: Infanrix hexa; Biological: Havrix; Biological: Varilrix
- Unprimed Group (Experimental): This group consisted of subjects between, and including, 64-68 months of age at the time of additional vaccination (primed subjects) or dose 1 (unprimed subjects), and for whom the investigator believed that their parents/guardians could and would comply with the requirements of the protocol. Subjects were not previously vaccinated with any pneumococcal vaccine and received 2 doses of Synflorix vaccine at 64-68 and 66-70 months of age (at Day 0 and Month 2).
  The Unprimed Group was added only in Year 4 of the study.
  Interventions: Biological: GSK1024805A

INTERVENTIONS:
Biological: GSK1024805A — No vaccination in this trial
  Other Names: Synflorix
  Arms: Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix; Synflorix + Infanrix + Havrix and/or Varilrix Group; Unprimed Group
Biological: Prevenar — No vaccination in this trial
  Arms: Prevenar + Infanrix + Havrix and/or Varilrix Group; Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Biological: Infanrix hexa — No vaccination in this trial
  Arms: Prevenar + Infanrix + Havrix and/or Varilrix Group; Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix; Synflorix + Infanrix + Havrix and/or Varilrix Group
Biological: Havrix — No vaccination in this trial
  Arms: Prevenar + Infanrix + Havrix and/or Varilrix Group; Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix; Synflorix + Infanrix + Havrix and/or Varilrix Group
Biological: Varilrix — No vaccination in this trial
  Arms: Prevenar + Infanrix + Havrix and/or Varilrix Group; Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix; Synflorix + Infanrix + Havrix and/or Varilrix Group

SUMMARY:
This protocol posting deals with objectives & outcome measures of the extension phase up to 48-50 months post booster vaccination, to assess long-term antibody persistence in children at around 30, 42 and 66 months of age, who received previously 4 doses of pneumococcal conjugate vaccine. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = 00307554). This Protocol posting has been updated in order to comply with the FDA AA (Sep 2007).

DETAILED DESCRIPTION:
This study consists in a serological follow-up study to evaluate persistence 12, 24 and 48 months after the booster vaccination study (107046). No study vaccines will be administered within this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 28-30 months of age at the time of first blood sampling.
* Subjects who previously participated in the 105553 and 107046 studies and who received a full four dose regimen of pneumococcal conjugate vaccine during the primary and booster studies.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Written informed consent, covering visits 1, 2 and 3, obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the blood sampling
* Administration of any additional pneumococcal vaccine since end of 107046 study.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the blood sampling.
* Administration of immunoglobulins and/or any blood products less than 6 months prior to blood sampling.
* Any confirmed or suspected immunosuppressive or immunodeficient condition since the end of the 107046 study, based on medical history and physical examination.

Ages: 28 Months to 32 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 524 (Actual)
Dates: Start 2008-03-03 (Actual); Primary Completion 2008-06-02 (Actual); Study Completion 2008-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=2213

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111345 (Mth 12) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primed groups included Synflorix vaccinated subjects in study 10PN-PD-DIT-007. The Unprimed Group, added only in Year 4,included subjects unprimed with any pneumococcal vaccine age-matched with primed groups. The study included 3 sub-studies (111345, 111346, 111347) corresponding to Year 1, 2 and 4 time points post Dose 1 in Study 10PN-PD-DIT-001.
Pre-assignment Details: At screening, subjects with previous participation in 10PN-PD-DIT-007 study were invited to join this study. Informed consent was obtained and signed from subjects' parents/guardians, check for inclusion/exclusion criteria and contraindications/precautions was performed, and medical history of subjects was collected.
Period: Follow-up Period: Year 1
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Started | 391 | 31 | 102 | 0
Completed | 391 | 31 | 102 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Follow-up Period: Year 2
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Started | 370 | 31 | 96 | 0
Completed | 370 | 31 | 96 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Follow-up Period: Year 4
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Started | 264 | 20 | 65 | 100
Completed | 263 | 19 | 64 | 100
Not Completed | 1 | 1 | 1 | 0
Not completed — Parents decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The demographic characteristics are presented separately for each Follow-up Period (Year 1, 2 and 4).
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group | Total
Number analyzed (Participants) | 391 | 31 | 102 | 100 | 624
Age, Continuous [Mean (Standard Deviation); unit: Months] — Data was presented for Follow-up Period: Year 1 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Months
    number analyzed (Participants) | 391 | 31 | 102 | 0 | 524
    (all) | 29.1 (0.88) | 29.0 (0.75) | 29.1 (0.81) |  | 29.1 (0.86)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Data was presented for Follow-up Period: Year 2 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Months
    number analyzed (Participants) | 370 | 31 | 96 | 0 | 497
    (all) | 41.1 (1.04) | 41.1 (1.09) | 41.2 (1.04) |  | 41.1 (1.04)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Data was presented for Follow-up Period: Year 4 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Months
    number analyzed (Participants) | 264 | 20 | 65 | 100 | 449
    (all) | 67.4 (0.84) | 67.1 (0.97) | 67.3 (0.89) | 65.4 (1.31) | 66.9 (1.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Data was presented for Follow-up Period Year 1 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    number analyzed (Participants) | 391 | 31 | 102 | 0 | 524
    Female | 203 | 14 | 52 |  | 269
    Male | 188 | 17 | 50 |  | 255
Sex: Female, Male [Count of Participants; unit: Participants] — Data was presented for Follow-up Period: Year 2 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    number analyzed (Participants) | 370 | 31 | 96 | 0 | 497
    Female | 192 | 14 | 50 |  | 256
    Male | 178 | 17 | 46 |  | 241
Sex: Female, Male [Count of Participants; unit: Participants] — Data was presented for Follow-up Period: Year 4 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    number analyzed (Participants) | 264 | 20 | 65 | 100 | 449
    Female | 139 | 10 | 35 | 53 | 237
    Male | 125 | 10 | 30 | 47 | 212
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data was presented for Follow-up Period: Year 1 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    White - caucasia/ european heritage: number analyzed (Participants) | 391 | 31 | 102 | 0 | 524
    White - caucasia/ european heritage | 386 | 31 | 102 | 0 | 519
    White arabic/ north african heritage: number analyzed (Participants) | 391 | 31 | 102 | 0 | 524
    White arabic/ north african heritage | 4 | 0 | 4 | 0 | 8
    Other, not specified: number analyzed (Participants) | 391 | 31 | 102 | 0 | 524
    Other, not specified | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data was presented for Follow-up Period: Year 2 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    number analyzed (Participants) | 370 | 31 | 96 | 0 | 497
    White - Caucasian / European heritage | 365 | 31 | 96 | 0 | 492
    White - Arabic / North African heritage | 4 | 0 | 0 | 0 | 4
    Other, not specified | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data was presented for Follow-up Period: Year 4 Population: Demographic characteristics data was presented for each Follow-up Period (Year 1, 2 and 4). Unprimed Group was added only in Year 4 of the study.
  Participants
    number analyzed (Participants) | 264 | 20 | 65 | 100 | 449
    White - Caucasian/ European heritage | 261 | 20 | 65 | 98 | 444
    White - Arabic/North African heritage | 3 | 0 | 0 | 0 | 3
    Asian - Central/South Asian heritage | 0 | 0 | 0 | 1 | 1
    Other, not specified | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-vaccine Pneumococcal Serotypes Antibody Concentrations Greater Than or Equal to (≥) the Cut-off [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Analysis was performed using the 22F-inhibition Enzyme-linked immunosorbent assay (ELISA), using 0.05 microgram per milliliter (µg/mL) as seropositivity cut off.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The According-To-Protocol (ATP) cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 389 | 31 | 102
Participants
  Anti-1 antibodies, Y1: number analyzed (Participants) | 387 | 29 | 102
  Anti-1 antibodies, Y1 | 372 | 7 | 99
  Anti-4 antibodies, Y1: number analyzed (Participants) | 387 | 31 | 102
  Anti-4 antibodies, Y1 | 384 | 31 | 102
  Anti-5 antibodies, Y1: number analyzed (Participants) | 387 | 30 | 101
  Anti-5 antibodies, Y1 | 386 | 19 | 101
  Anti-6B antibodies, Y1 | 384 | 31 | 100
  Anti-7F antibodies, Y1: number analyzed (Participants) | 387 | 31 | 102
  Anti-7F antibodies, Y1 | 387 | 17 | 102
  Anti-9V antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-9V antibodies, Y1 | 388 | 17 | 102
  Anti-14 antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-14 antibodies, Y1 | 387 | 31 | 102
  Anti-18C antibodies, Y1: number analyzed (Participants) | 384 | 31 | 102
  Anti-18C antibodies, Y1 | 384 | 31 | 102
  Anti-19F antibodies, Y1: number analyzed (Participants) | 387 | 31 | 102
  Anti-19F antibodies, Y1 | 387 | 31 | 102
  Anti-23F antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-23F antibodies, Y1 | 386 | 31 | 102

2. Primary Outcome: Number of Subjects With Anti-vaccine Pneumococcal Serotypes Antibody Concentrations ≥ the Cut-off [Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Analysis was performed using the 22F-inhibition Enzyme -linked immunosorbent assay (ELISA), using 0.05 μg/mL as seropositivity cut off.
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The ATP cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 30 | 96
Participants
  Anti-1 antibodies, Y2: number analyzed (Participants) | 367 | 29 | 96
  Anti-1 antibodies, Y2 | 354 | 18 | 90
  Anti-4 antibodies, Y2 | 356 | 30 | 96
  Anti-5 antibodies, Y2: number analyzed (Participants) | 368 | 29 | 95
  Anti-5 antibodies, Y2 | 362 | 21 | 95
  Anti-6B antibodies, Y2 | 355 | 30 | 95
  Anti-7F antibodies, Y2 | 367 | 19 | 95
  Anti-9V antibodies, Y2 | 362 | 30 | 96
  Anti-14 antibodies, Y2 | 367 | 30 | 96
  Anti-18C antibodies, Y2 | 365 | 30 | 96
  Anti-19F antibodies, Y2: number analyzed (Participants) | 368 | 30 | 95
  Anti-19F antibodies, Y2 | 368 | 30 | 95
  Anti-23F antibodies, Y2 | 357 | 30 | 95

3. Primary Outcome: Number of Subjects With Anti-vaccine Pneumococcal Serotypes Antibody Concentrations ≥ the Cut-off [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Analysis was performed using the 22F-inhibition Enzyme-linked immunosorbent assay (ELISA), using 0.05 μg/mL as seropositivity cut off.
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The ATP cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 264 | 19 | 75
Participants
  Anti-1 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-1 antibodies, Y4 | 238 | 14 | 71
  Anti-4 antibodies, Y4: number analyzed (Participants) | 263 | 18 | 74
  Anti-4 antibodies, Y4 | 238 | 18 | 72
  Anti-5 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-5 antibodies, Y4 | 257 | 19 | 73
  Anti-6B antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-6B antibodies, Y4 | 258 | 19 | 74
  Anti-7F antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-7F antibodies, Y4 | 260 | 13 | 73
  Anti-9V antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-9V antibodies, Y4 | 255 | 19 | 75
  Anti-14 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-14 antibodies, Y4 | 263 | 19 | 75
  Anti-18C antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-18C antibodies, Y4 | 256 | 19 | 73
  Anti-19F antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-19F antibodies, Y4 | 260 | 19 | 75
  Anti-23F antibodies, Y4: number analyzed (Participants) | 262 | 19 | 75
  Anti-23F antibodies, Y4 | 254 | 19 | 74

4. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes [Follow-Up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: Pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Antibody concentrations against pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micro grams per milliliter (µg/mL).The seropositivity cut-off for the assay was ≥ 0.05 µg/mL.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The ATP cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 1.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 389 | 31 | 102
µg/mL
  Anti-1 antibodies, Y1: number analyzed (Participants) | 387 | 29 | 102
  Anti-1 antibodies, Y1 | 0.29 [0.27 to 0.32] | 0.04 [0.03 to 0.06] | 0.26 [0.21 to 0.31]
  Anti-4 antibodies, Y1: number analyzed (Participants) | 387 | 31 | 102
  Anti-4 antibodies, Y1 | 0.5 [0.45 to 0.55] | 0.59 [0.46 to 0.75] | 1.01 [0.84 to 1.21]
  Anti-5 antibodies, Y1: number analyzed (Participants) | 387 | 30 | 101
  Anti-5 antibodies, Y1 | 0.59 [0.54 to 0.65] | 0.07 [0.05 to 0.11] | 0.42 [0.35 to 0.52]
  Anti-6B antibodies, Y1 | 0.52 [0.45 to 0.6] | 0.98 [0.63 to 1.53] | 0.54 [0.42 to 0.69]
  Anti-7F antibodies, Y1: number analyzed (Participants) | 387 | 31 | 102
  Anti-7F antibodies, Y1 | 0.71 [0.66 to 0.77] | 0.08 [0.05 to 0.13] | 0.83 [0.7 to 0.99]
  Anti-9V antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-9V antibodies, Y1 | 0.79 [0.71 to 0.89] | 0.93 [0.7 to 1.22] | 0.58 [0.49 to 0.68]
  Anti-14 antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-14 antibodies, Y1 | 1.27 [1.12 to 1.44] | 1.79 [1.29 to 2.48] | 1.47 [1.17 to 1.85]
  Anti-18C antibodies, Y1: number analyzed (Participants) | 384 | 31 | 102
  Anti-18C antibodies, Y1 | 0.88 [0.81 to 0.96] | 0.91 [0.71 to 1.16] | 0.82 [0.69 to 0.98]
  Anti-19F antibodies, Y1: number analyzed (Participants) | 387 | 30 | 102
  Anti-19F antibodies, Y1 | 1.43 [1.27 to 1.6] | 0.83 [0.47 to 1.45] | 1.51 [1.19 to 1.92]
  Anti-23F antibodies, Y1: number analyzed (Participants) | 388 | 31 | 102
  Anti-23F antibodies, Y1 | 0.61 [0.54 to 0.69] | 1.18 [0.84 to 1.68] | 0.7 [0.56 to 0.88]

5. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes [Follow-Up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: Pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Antibody concentrations against pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micro grams per milliliter (µg/mL). The seropositivity cut-off for the assay was ≥ 0.05 µg/mL.
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 30 | 96
µg/mL
  Anti-1 antibodies, Y2: number analyzed (Participants) | 367 | 29 | 96
  Anti-1 antibodies, Y2 | 0.19 [0.17 to 0.21] | 0.07 [0.05 to 0.1] | 0.17 [0.14 to 0.2]
  Anti-4 antibodies, Y2 | 0.27 [0.24 to 0.3] | 0.3 [0.24 to 0.38] | 0.52 [0.43 to 0.64]
  Anti-5 antibodies, Y2: number analyzed (Participants) | 368 | 29 | 95
  Anti-5 antibodies, Y2 | 0.41 [0.37 to 0.45] | 0.09 [0.06 to 0.13] | 0.33 [0.27 to 0.41]
  Anti-6B antibodies, Y2 | 0.7 [0.58 to 0.83] | 0.99 [0.57 to 1.71] | 0.9 [0.63 to 1.29]
  Anti-7F antibodies, Y2 | 0.53 [0.48 to 0.58] | 0.1 [0.06 to 0.16] | 0.59 [0.49 to 0.71]
  Anti-9V antibodies, Y2 | 0.64 [0.54 to 0.75] | 0.61 [0.37 to 1] | 0.5 [0.37 to 0.68]
  Anti-14 antibodies, Y2 | 1.73 [1.48 to 2.02] | 1.94 [1.12 to 3.36] | 1.7 [1.25 to 2.31]
  Anti-18C antibodies, Y2 | 0.54 [0.48 to 0.62] | 0.59 [0.39 to 0.88] | 0.48 [0.38 to 0.59]
  Anti-19F antibodies, Y2: number analyzed (Participants) | 368 | 30 | 95
  Anti-19F antibodies, Y2 | 2.16 [1.77 to 2.65] | 0.99 [0.51 to 1.91] | 2.41 [1.67 to 3.46]
  Anti-23F antibodies, Y2 | 0.68 [0.56 to 0.82] | 1.24 [0.83 to 1.85] | 0.64 [0.48 to 0.86]

6. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: Pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Antibody concentrations against pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micro grams per milliliter (µg/mL). The seropositivity cut-off for the assay was ≥ 0.05 μg/mL.
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PDDIT- 007)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 264 | 19 | 75
μg/mL
  Anti-1 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-1 antibodies, Y4 | 0.2 [0.17 to 0.24] | 0.17 [0.07 to 0.43] | 0.23 [0.17 to 0.32]
  Anti-4 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-4 antibodies, Y4 | 0.19 [0.16 to 0.22] | 0.23 [0.12 to 0.41] | 0.31 [0.25 to 0.38]
  Anti-5 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-5 antibodies, Y4 | 0.36 [0.31 to 0.4] | 0.19 [0.1 to 0.35] | 0.35 [0.28 to 0.43]
  Anti-6B antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-6B antibodies, Y4 | 1.3 [1.1 to 1.55] | 1.19 [0.68 to 2.07] | 0.97 [0.74 to 1.27]
  Anti-7F antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-7F antibodies, Y4 | 0.44 [0.38 to 0.52] | 0.16 [0.08 to 0.36] | 0.49 [0.37 to 0.65]
  Anti-9V antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-9V antibodies, Y4 | 1.17 [0.92 to 1.47] | 1.19 [0.43 to 3.27] | 0.67 [0.46 to 0.99]
  Anti-14 antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-14 antibodies, Y4 | 3.66 [3.01 to 4.45] | 2.57 [1.22 to 5.42] | 2.94 [2.11 to 4.12]
  Anti-18C antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-18C antibodies, Y4 | 0.7 [0.58 to 0.84] | 0.87 [0.4 to 1.88] | 0.63 [0.45 to 0.89]
  Anti-19F antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-19F antibodies, Y4 | 4.17 [3.4 to 5.1] | 4.74 [2.24 to 10] | 4.05 [3.03 to 5.41]
  Anti-23F antibodies, Y4: number analyzed (Participants) | 262 | 19 | 75
  Anti-23F antibodies, Y4 | 1.57 [1.26 to 1.96] | 1.64 [1.15 to 2.34] | 1.12 [0.79 to 1.58]

7. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: Anti-pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F . Antibody concentrations against pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micro grams per milliliter (µg/mL). The seropositivity cut-off for the assay was ≥ 0.05 μg/mL.
Time Frame: For primed groups: At Month 48+7 days after additional dose (D7);For unprimed group: at Day 0 (D0) (Pre-vaccination [PRE]), at Day 7 (D7) post dose 1 (of the 2-dose catch-up vaccination) and at Month 3 (M3) post dose 2 (of the 2-dose catch-up vaccination)
Population: The ATP cohort for immunogenicity included all evaluable subjects for whom assay results were available for antibodies against at least one vaccine antigen component for blood samples taken 7 days after additional dose (primed subjects) or at pre-vaccination, 7 days post-dose 1, and 1-month post-dose 2 catch-up vaccination (unprimed subjects).
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 210 | 14 | 55 | 98
μg/mL
  Anti-1 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-1 antibodies, PRE |  |  |  | 0.1 [0.08 to 0.13]
  Anti-1 antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-1 antibodies, D7 | 5.36 [4.54 to 6.33] | 3.04 [1.22 to 7.56] | 5 [3.72 to 6.71] | 1.35 [1.08 to 1.69]
  Anti-1 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-1 antibodies, M3 |  |  |  | 2.39 [2.06 to 2.78]
  Anti-4 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-4 antibodies, PRE |  |  |  | 0.04 [0.03 to 0.05]
  Anti-4 antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-4 antibodies, D7 | 12.11 [10.08 to 14.54] | 10.45 [6.49 to 16.81] | 7.13 [5.18 to 9.82] | 4.74 [3.77 to 5.95]
  Anti-4 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-4 antibodies, M3 |  |  |  | 7.32 [6.7 to 8]
  Anti-5 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-5 antibodies, PRE |  |  |  | 0.1 [0.08 to 0.12]
  Anti-5 antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-5 antibodies, D7 | 6.23 [5.19 to 7.49] | 3.24 [1.44 to 7.29] | 8.15 [5.71 to 11.63] | 1.2 [0.97 to 1.49]
  Anti-5 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-5 antibodies, M3 |  |  |  | 3.1 [2.7 to 3.55]
  Anti-6B antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-6B antibodies, PRE |  |  |  | 0.21 [0.15 to 0.29]
  Anti-6B antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 97
  Anti-6B antibodies, D7 | 3.68 [3.16 to 4.29] | 2.85 [1.89 to 4.3] | 2.15 [1.62 to 2.85] | 0.53 [0.4 to 0.71]
  Anti-6B antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-6B antibodies, M3 |  |  |  | 1.25 [1.01 to 1.54]
  Anti-7F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-7F antibodies, PRE |  |  |  | 0.12 [0.09 to 0.16]
  Anti-7F antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-7F antibodies, D7 | 7.16 [6.11 to 8.39] | 3.26 [1.67 to 6.35] | 7.57 [5.84 to 9.81] | 1.67 [1.33 to 2.09]
  Anti-7F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-7F antibodies, M3 |  |  |  | 4.55 [3.93 to 5.26]
  Anti-9V antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-9V antibodies, PRE |  |  |  | 0.19 [0.12 to 0.28]
  Anti-9V antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-9V antibodies, D7 | 9.94 [8.59 to 11.51] | 9 [5.49 to 14.77] | 5.32 [4.08 to 6.94] | 0.9 [0.66 to 1.23]
  Anti-9V antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-9V antibodies, M3 |  |  |  | 2.2 [1.85 to 2.62]
  Anti-14 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-14 antibodies, PRE |  |  |  | 0.58 [0.38 to 0.87]
  Anti-14 antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-14 antibodies, D7 | 19.38 [16.74 to 22.43] | 13.26 [6.91 to 25.43] | 18.61 [14.23 to 24.34] | 1.72 [1.2 to 2.46]
  Anti-14 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-14 antibodies, M3 |  |  |  | 7.81 [6.34 to 9.63]
  Anti-18C antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-18C antibodies, PRE |  |  |  | 0.1 [0.07 to 0.15]
  Anti-18C antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-18C antibodies, D7 | 15.51 [13.06 to 18.43] | 19.71 [11.87 to 32.74] | 13.34 [9.34 to 19.05] | 2.26 [1.66 to 3.09]
  Anti-18C antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-18C antibodies, M3 |  |  |  | 13.21 [11.44 to 15.25]
  Anti-19F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-19F antibodies, PRE |  |  |  | 0.6 [0.4 to 0.89]
  Anti-19F antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-19F antibodies, D7 | 11.63 [10 to 13.51] | 16.44 [10.68 to 25.29] | 8.09 [6.29 to 10.42] | 5.12 [3.97 to 6.62]
  Anti-19F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-19F antibodies, M3 |  |  |  | 15.47 [13.08 to 18.29]
  Anti-23F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-23F antibodies, PRE |  |  |  | 0.1 [0.07 to 0.14]
  Anti-23F antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-23F antibodies, D7 | 6.5 [5.61 to 7.53] | 9.34 [5.62 to 15.54] | 4.7 [3.43 to 6.45] | 0.42 [0.3 to 0.59]
  Anti-23F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-23F antibodies, M3 |  |  |  | 1.63 [1.32 to 2.01]

8. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes [Follow-Up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: Pneumococcal serotypes assessed were OPA-1, OPA-4, OPA-5, OPA-6B, OPA-7F, OPA-9V, OPA-14, OPA-18C, OPA-19F and OPA-23F. The seropositivity cut-off for the assay was ≥ 8. Opsonophagocytic activity was expressed as Geometric Mean Antibody Titers (GMT).
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 359 | 27 | 94
Titer
  Anti-1 OPA Titers, Y1: number analyzed (Participants) | 354 | 27 | 92
  Anti-1 OPA Titers, Y1 | 16.2 [13.8 to 19] | 4.8 [3.6 to 6.4] | 7.3 [5.9 to 9]
  Anti-4 OPA Titers, Y1: number analyzed (Participants) | 340 | 26 | 86
  Anti-4 OPA Titers, Y1 | 59.8 [45.7 to 78.3] | 192.9 [82.4 to 452] | 88.9 [54.6 to 144.6]
  Anti-5 OPA Titers, Y1: number analyzed (Participants) | 335 | 27 | 89
  Anti-5 OPA Titers, Y1 | 24.2 [20.8 to 28.2] | 5.1 [3.6 to 7.4] | 11.2 [8.7 to 14.3]
  Anti-6B OPA Titers, Y1: number analyzed (Participants) | 354 | 25 | 88
  Anti-6B OPA Titers, Y1 | 35.5 [26.5 to 47.5] | 476.9 [175.3 to 1298] | 44.7 [24 to 83.3]
  Anti-7F OPA Titers, Y1: number analyzed (Participants) | 346 | 25 | 89
  Anti-7F OPA Titers, Y1 | 1855.7 [1644.4 to 2094.1] | 350.4 [121.8 to 1008] | 1617.2 [1152.9 to 2268.3]
  Anti-9V OPA Titers, Y1: number analyzed (Participants) | 352 | 26 | 94
  Anti-9V OPA Titers, Y1 | 791.5 [701.8 to 892.8] | 1240.7 [829.4 to 1855.9] | 370.5 [281.8 to 487.2]
  Anti-14 OPA Titers, Y1: number analyzed (Participants) | 343 | 25 | 91
  Anti-14 OPA Titers, Y1 | 551.9 [486.5 to 626.2] | 607.3 [385.3 to 957.1] | 456.6 [361.1 to 577.3]
  Anti-18C OPA Titers, Y1: number analyzed (Participants) | 319 | 24 | 84
  Anti-18C OPA Titers, Y1 | 23.5 [18.6 to 29.8] | 15.5 [6.1 to 39.2] | 10.4 [7.1 to 15.4]
  Anti-19F OPA Titers, Y1 | 53.4 [44.7 to 63.9] | 35.4 [15.9 to 78.6] | 58 [41.6 to 80.7]
  Anti-23F OPA Titers, Y1: number analyzed (Participants) | 336 | 27 | 93
  Anti-23F OPA Titers, Y1 | 784.9 [625.4 to 985] | 3013.1 [1349.5 to 6727.2] | 552.3 [362.1 to 842.5]

9. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes [Follow-Up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: as for outcome 8
Time Frame: At Year 2 (Y2) (post booster vaccination administrated in study 10PN-PD-DIT-007)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 354 | 27 | 92
Titer
  Anti-1 OPA Titers, Y2 | 8.4 [7.3 to 9.7] | 4 [4 to 4] | 6.3 [4.9 to 8]
  Anti-4 OPA Titers, Y2: number analyzed (Participants) | 335 | 27 | 84
  Anti-4 OPA Titers, Y2 | 29 [22.1 to 38] | 33.5 [11.9 to 94.6] | 39.3 [23.7 to 65.2]
  Anti-5 OPA Titers, Y2: number analyzed (Participants) | 351 | 27 | 91
  Anti-5 OPA Titers, Y2 | 11.4 [10 to 13] | 4.3 [3.9 to 4.7] | 7.4 [6 to 9.1]
  Anti-6B OPA Titers, Y2: number analyzed (Participants) | 342 | 27 | 88
  Anti-6B OPA Titers, Y2 | 167.2 [124.1 to 225.2] | 526.1 [210.5 to 1314.4] | 213.7 [117.8 to 387.6]
  Anti-7F OPA Titers, Y2: number analyzed (Participants) | 350 | 27 | 91
  Anti-7F OPA Titers, Y2 | 1488.7 [1358.3 to 1631.6] | 1068.3 [619.5 to 1842.4] | 1387.8 [1096.2 to 1756.9]
  Anti-9V OPA Titers, Y2: number analyzed (Participants) | 349 | 27 | 92
  Anti-9V OPA Titers, Y2 | 648.5 [570 to 737.7] | 730.4 [457.7 to 1165.7] | 391 [279.2 to 547.5]
  Anti-14 OPA Titers, Y2: number analyzed (Participants) | 341 | 25 | 90
  Anti-14 OPA Titers, Y2 | 660.2 [567.2 to 768.4] | 651 [348.6 to 1215.5] | 534.4 [381.6 to 748.4]
  Anti-18C OPA Titers, Y2: number analyzed (Participants) | 325 | 27 | 83
  Anti-18C OPA Titers, Y2 | 34.9 [26.6 to 45.7] | 34.8 [11.7 to 103.2] | 17.7 [10.7 to 29.2]
  Anti-19F OPA Titers, Y2: number analyzed (Participants) | 349 | 27 | 92
  Anti-19F OPA Titers, Y2 | 78.1 [60.9 to 100.2] | 49.2 [21.2 to 113.9] | 105.4 [65.8 to 168.7]
  Anti-23F OPA Titers, Y2: number analyzed (Participants) | 342 | 26 | 91
  Anti-23F OPA Titers, Y2 | 632 [483 to 827] | 1923 [952.2 to 3883.7] | 435 [250.5 to 755.5]

10. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: Pneumococcal serotypes assessed were pneumococcal serotypes OPA-1, OPA-4, OPA-5, OPA-6B, OPA-7F, OPA-9V, OPA-14, OPA-18C, OPA-19F and OPA-23F. The seropositivity cut-off for the assay was ≥ 8. Opsonophagocytic activity was expressed as Geometric Mean Antibody Titers (GMT).
Time Frame: At Year 4 (Y4) (post booster vaccination administrated in study 10PN-PD-DIT-007)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 253 | 16 | 72
Titer
  Anti-1 OPA Titers, Y4: number analyzed (Participants) | 250 | 16 | 72
  Anti-1 OPA Titers, Y4 | 8.8 [7.1 to 10.9] | 4.6 [3.4 to 6.4] | 8.9 [5.9 to 13.2]
  Anti-4 OPA Titers, Y4: number analyzed (Participants) | 232 | 16 | 63
  Anti-4 OPA Titers, Y4 | 37.9 [27.2 to 52.8] | 62.2 [13.6 to 284.7] | 50.7 [26.5 to 97]
  Anti-5 OPA Titers, Y4: number analyzed (Participants) | 243 | 15 | 68
  Anti-5 OPA Titers, Y4 | 7.7 [6.8 to 8.9] | 5.3 [3.5 to 8.1] | 5.5 [4.5 to 6.6]
  Anti-6B OPA Titers, Y4: number analyzed (Participants) | 250 | 16 | 68
  Anti-6B OPA Titers, Y4 | 875.7 [658.7 to 1164.3] | 978.3 [395.3 to 2421.3] | 716.4 [417.4 to 1229.7]
  Anti-7F OPA Titers, Y4: number analyzed (Participants) | 249 | 15 | 71
  Anti-7F OPA Titers, Y4 | 1693.1 [1489.3 to 1924.8] | 965.8 [666.8 to 1398.9] | 1602.1 [1286.9 to 1994.5]
  Anti-9V OPA Titers, Y4: number analyzed (Participants) | 250 | 15 | 70
  Anti-9V OPA Titers, Y4 | 747.4 [624.9 to 894.1] | 563.8 [220.2 to 1444] | 558.6 [403 to 774.2]
  Anti-14 OPA Titers, Y4: number analyzed (Participants) | 250 | 15 | 71
  Anti-14 OPA Titers, Y4 | 1139.8 [961.9 to 1350.5] | 687.9 [267.8 to 1767.4] | 849.4 [645.4 to 1117.8]
  Anti-18C OPA Titers, Y4: number analyzed (Participants) | 226 | 16 | 63
  Anti-18C OPA Titers, Y4 | 46.4 [33.3 to 64.5] | 35.3 [8.8 to 142.5] | 26.6 [14.3 to 49.3]
  Anti-19F OPA Titers, Y4: number analyzed (Participants) | 247 | 16 | 69
  Anti-19F OPA Titers, Y4 | 151.7 [115.9 to 198.4] | 178.8 [64.6 to 495.1] | 129.3 [83.1 to 201.4]
  Anti-23F OPA Titers, Y4: number analyzed (Participants) | 239 | 15 | 65
  Anti-23F OPA Titers, Y4 | 1518.4 [1107.9 to 2080.9] | 3366.1 [1599.2 to 7085.1] | 1146.2 [596.8 to 2201.3]

11. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 204 | 13 | 54 | 96
Titers
  Anti-1 OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-1 OPA Titers, PRE |  |  |  | 5 [4.2 to 5.9]
  Anti-1 OPA Titers, D7: number analyzed (Participants) | 197 | 13 | 50 | 92
  Anti-1 OPA Titers, D7 | 2920.8 [2353.5 to 3624.7] | 1331 [586.7 to 3019.5] | 1816.1 [1090 to 3025.8] | 605 [462.7 to 791.2]
  Anti-1 OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-1 OPA Titers, M3 |  |  |  | 128.3 [97.3 to 169.1]
  Anti-4 OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 81
  Anti-4 OPA Titers, PRE |  |  |  | 11.5 [7.2 to 18.3]
  Anti-4 OPA Titers, D7: number analyzed (Participants) | 196 | 13 | 51 | 93
  Anti-4 OPA Titers, D7 | 23633.7 [19118.5 to 29215.3] | 10650.3 [3969.2 to 28577.6] | 8592.8 [5609.3 to 13163.1] | 18262.1 [15571.6 to 21417.4]
  Anti-4 OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-4 OPA Titers, M3 |  |  |  | 4451.3 [3962.4 to 5000.6]
  Anti-5 OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 91
  Anti-5 OPA Titers, PRE |  |  |  | 4.9 [4.3 to 5.7]
  Anti-5 OPA Titers, D7: number analyzed (Participants) | 193 | 13 | 48 | 91
  Anti-5 OPA Titers, D7 | 822.3 [662.7 to 1020.3] | 375.6 [217.4 to 648.9] | 683.6 [428.6 to 1090.2] | 295.6 [219.4 to 398.3]
  Anti-5 OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-5 OPA Titers, M3 |  |  |  | 93.2 [73.7 to 117.8]
  Anti-6B OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 79
  Anti-6B OPA Titers, PRE |  |  |  | 70.7 [33.5 to 149.2]
  Anti-6B OPA Titers, D7: number analyzed (Participants) | 198 | 13 | 50 | 93
  Anti-6B OPA Titers, D7 | 3513.1 [2858.1 to 4318.1] | 3566.6 [2446.1 to 5200.3] | 1590.5 [942.8 to 2683.3] | 1971.4 [1238 to 3139.2]
  Anti-6B OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-6B OPA Titers, M3 |  |  |  | 2536.9 [2014.1 to 3195.5]
  Anti-7F OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 74
  Anti-7F OPA Titers, PRE |  |  |  | 1368.2 [849.6 to 2185.8]
  Anti-7F OPA Titers, D7: number analyzed (Participants) | 199 | 13 | 50 | 93
  Anti-7F OPA Titers, D7 | 25196.4 [21149.5 to 30017.6] | 17828.8 [10270.4 to 30949.7] | 13098.6 [9715.5 to 17659.8] | 19243.4 [15701.4 to 23584.5]
  Anti-7F OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 93
  Anti-7F OPA Titers, M3 |  |  |  | 9692 [8299.3 to 11318.4]
  Anti-9V OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 87
  Anti-9V OPA Titers, PRE |  |  |  | 398.2 [253.8 to 624.9]
  Anti-9V OPA Titers, D7: number analyzed (Participants) | 201 | 13 | 51 | 93
  Anti-9V OPA Titers, D7 | 9419.4 [7586 to 11695.9] | 12234.7 [8280.5 to 18077.3] | 7730.3 [5361.8 to 11145.2] | 8322.7 [6605.7 to 10486.1]
  Anti-9V OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-9V OPA Titers, M3 |  |  |  | 6456.1 [5458.1 to 7636.6]
  Anti-14 OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 83
  Anti-14 OPA Titers, PRE |  |  |  | 586.5 [439 to 783.6]
  Anti-14 OPA Titers, D7: number analyzed (Participants) | 197 | 13 | 51 | 94
  Anti-14 OPA Titers, D7 | 8572.3 [7145.4 to 10284.3] | 4192.8 [2218.6 to 7923.7] | 6883.1 [5057.3 to 9368] | 4678.2 [3788 to 5777.5]
  Anti-14 OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-14 OPA Titers, M3 |  |  |  | 4891.1 [4178.8 to 5724.8]
  Anti-18C OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 89
  Anti-18C OPA Titers, PRE |  |  |  | 5.3 [4.2 to 6.6]
  Anti-18C OPA Titers, D7: number analyzed (Participants) | 194 | 13 | 50 | 92
  Anti-18C OPA Titers, D7 | 3378.9 [2652.2 to 4304.8] | 3478.6 [1788.5 to 6765.8] | 1663.2 [970.5 to 2850.2] | 2503.1 [1692.6 to 3701.6]
  Anti-18C OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-18C OPA Titers, M3 |  |  |  | 2255.9 [1876.9 to 2711.4]
  Anti-19F OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-19F OPA Titers, PRE |  |  |  | 12 [8.3 to 17.5]
  Anti-19F OPA Titers, D7: number analyzed (Participants) | 196 | 13 | 50 | 93
  Anti-19F OPA Titers, D7 | 1346.4 [1068.6 to 1696.5] | 2340.4 [654.8 to 8365.2] | 662.3 [430 to 1020.1] | 700.2 [456.1 to 1074.9]
  Anti-19F OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 93
  Anti-19F OPA Titers, M3 |  |  |  | 1437.7 [1146.9 to 1802.3]
  Anti-23F OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 83
  Anti-23F OPA Titers, PRE |  |  |  | 176.4 [83.4 to 373.2]
  Anti-23F OPA Titers, D7: number analyzed (Participants) | 199 | 13 | 50 | 96
  Anti-23F OPA Titers, D7 | 8700.4 [7021.7 to 10780.5] | 11341.1 [5374.6 to 23931] | 7871.9 [4965.3 to 12480.1] | 6813.9 [5249.5 to 8844.6]
  Anti-23F OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-23F OPA Titers, M3 |  |  |  | 5586.1 [4666.1 to 6687.5]

12. Secondary Outcome: Antibody Concentrations Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and - 19A) [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: The seropositivity cut-off for the assay was ≥ 0.05 μg/mL. Antibody concentrations against 6A and 19A pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micrograms per milliliter (µg/mL).
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 390 | 31 | 102
μg/mL
  Anti-6A antibodies, Y1 | 0.28 [0.24 to 0.32] | 0.44 [0.28 to 0.7] | 0.27 [0.21 to 0.36]
  Anti-19A antibodies, Y1 | 0.28 [0.25 to 0.32] | 0.21 [0.13 to 0.33] | 0.23 [0.17 to 0.3]

13. Secondary Outcome: Antibody Concentrations Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and - 19A) - Follow-Up Period: Persistence Analysis in Year 2 (111346 Sub-study)
Description: as for outcome 12
Time Frame: At Year 2 (Y2) (post booster vaccination administrated in study 10PN-PDDIT- 007)
Population: The analysis was performed on the ATP cohort for persistence, which included all subjects from the total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results were available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 2.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 30 | 96
μg/mL
  Anti-6A antibodies, Y2 | 0.33 [0.28 to 0.4] | 0.57 [0.3 to 1.11] | 0.4 [0.27 to 0.58]
  Anti-19A antibodies, Y2 | 0.37 [0.31 to 0.44] | 0.25 [0.14 to 0.44] | 0.35 [0.25 to 0.5]

14. Secondary Outcome: Antibody Concentrations Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and - 19A) [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: Antibody concentrations against 6A and 19A pneumococcal serotypes were determined as Geometric Mean Antibody Concentrations (GMC) and expressed as micro grams per milliliter (µg/mL). The seropositivity cut-off for the assay was ≥ 0.05 μg/mL.
Time Frame: At Year 4 (Y4) (post booster vaccination administrated in study 10PN-PD-DIT- 007)
Population: The analysis was a persistence analysis performed on the evaluable subjects enrolled in the applicable Year 4 Persistence and Immunological Memory 111347 Study, for whom assay results were available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 4.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 264 | 19 | 75
μg/mL
  Anti-6A antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-6A antibodies, Y4 | 0.92 [0.77 to 1.1] | 0.69 [0.34 to 1.38] | 0.75 [0.55 to 1.03]
  Anti-19A antibodies, Y4: number analyzed (Participants) | 263 | 19 | 75
  Anti-19A antibodies, Y4 | 1.3 [1.07 to 1.59] | 1.08 [0.5 to 2.33] | 1.14 [0.77 to 1.68]

15. Secondary Outcome: Antibody Concentrations Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and 19A) [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 14
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 210 | 14 | 55 | 98
μg/mL
  Anti-6A antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-6A antibodies, PRE |  |  |  | 0.2 [0.15 to 0.27]
  Anti-6A antibodies, D7: number analyzed (Participants) | 208 | 14 | 55 | 98
  Anti-6A antibodies, D7 | 2.2 [1.85 to 2.6] | 1.67 [1 to 2.8] | 1.33 [0.96 to 1.83] | 0.44 [0.33 to 0.58]
  Anti-6A antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-6A antibodies, M3 |  |  |  | 0.92 [0.73 to 1.16]
  Anti-19A antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-19A antibodies, PRE |  |  |  | 0.44 [0.32 to 0.6]
  Anti-19A antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 98
  Anti-19A antibodies, D7 | 2.79 [2.33 to 3.35] | 2.44 [1.2 to 4.96] | 1.72 [1.14 to 2.61] | 1.1 [0.84 to 1.45]
  Anti-19A antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-19A antibodies, M3 |  |  |  | 2.39 [1.9 to 3.01]

16. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Crossreactive Pneumococcal Serotypes 6A and 19 A [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: Opsonophagocytic activity were assessed for pneumococcal serotypes 6A and 19A (OPA-6A and OPA-19A). The seropositivity cut-off for the assay was ≥ 8. Opsonophagocytic activity was expressed as Geometric Mean Antibody Titers (GMT).
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 352 | 26 | 93
Titers
  Anti-6A OPA Titers, Y1: number analyzed (Participants) | 323 | 25 | 75
  Anti-6A OPA Titers, Y1 | 59 [45.9 to 76] | 610.2 [317.7 to 1171.9] | 46.6 [28.3 to 76.8]
  Anti-19A OPA Titers, Y1: number analyzed (Participants) | 155 | 26 | 93
  Anti-19A OPA Titers, Y1 | 6 [5.2 to 6.8] | 5.9 [3.7 to 9.5] | 5.5 [4.5 to 6.8]

17. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Crossreactive Pneumococcal Serotypes 6A and 19 A [Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: as for outcome 16
Time Frame: At Year 2 (Y2) (post booster vaccination administrated in study 10PN-PD-DIT-007)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 351 | 27 | 91
Titers
  Anti-6A OPA Titers, Y2: number analyzed (Participants) | 314 | 25 | 82
  Anti-6A OPA Titers, Y2 | 121.8 [95.2 to 156] | 356.5 [134.6 to 944.6] | 133.7 [81.8 to 218.7]
  Anti-19A OPA Titers, Y2 | 12.8 [10.4 to 15.7] | 10.9 [5.2 to 22.8] | 11.1 [7.6 to 16.2]

18. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Crossreactive Pneumococcal Serotypes 6A and 19 A [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 16
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The analysis was a persistence analysis performed on the evaluable subjects enrolled in the applicable Year 4 Persistence and Immunological Memory 111347 Study for whom assay results were available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 251 | 16 | 71
Titers
  Anti-6A OPA Titers, Y4: number analyzed (Participants) | 231 | 14 | 66
  Anti-6A OPA Titers, Y4 | 213.5 [165.4 to 275.7] | 227.8 [72.1 to 720] | 153.5 [90.5 to 260.2]
  Anti-19A OPA Titers, Y4: number analyzed (Participants) | 246 | 15 | 68
  Anti-19A OPA Titers, Y4 | 31.2 [23.6 to 41.3] | 14.3 [5.6 to 36.8] | 21.8 [13.3 to 35.7]

19. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 6A and 19A [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 16
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 201 | 13 | 50 | 92
Titers
  Anti-6A OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 82
  Anti-6A OPA Titers, PRE |  |  |  | 102.6 [61.5 to 171.2]
  Anti-6A OPA Titers, D7: number analyzed (Participants) | 189 | 12 | 49 | 90
  Anti-6A OPA Titers, D7 | 1217.7 [957.8 to 1548.2] | 1490.2 [681.6 to 3257.8] | 467.7 [293.8 to 744.5] | 826.5 [593.9 to 1150.2]
  Anti-6A OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 91
  Anti-6A OPA Titers, M3 |  |  |  | 943.4 [691.3 to 1287.4]
  Anti-19A OPA Titers, PRE: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-19A OPA Titers, PRE |  |  |  | 9.9 [7 to 13.8]
  Anti-19A OPA Titers, D7: number analyzed (Participants) | 194 | 13 | 48 | 90
  Anti-19A OPA Titers, D7 | 467 [335 to 651.1] | 437.6 [81.3 to 2356.3] | 106.1 [54.1 to 208.3] | 431.2 [269.4 to 689.9]
  Anti-19A OPA Titers, M3: number analyzed (Participants) | 0 | 0 | 0 | 91
  Anti-19A OPA Titers, M3 |  |  |  | 376.4 [256.3 to 552.6]

20. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD) - Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)
Description: Anti-protein D (Anti-PD) antibody concentrations by Enzyme-Linked Immunosorbent Assay (ELISA) were calculated, expressed as geometric mean concentrations (GMCs) in ELISA unit per milli-liter (EL.U/mL) and tabulated. The seropositivity cut-off for the assay was ≥ 100 EL.U/mL.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 390 | 30 | 102
EL.U/mL | 822.1 [731.5 to 923.9] | 93.9 [66.6 to 132.3] | 193.6 [155.9 to 240.4]

21. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD) - Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)
Description: as for outcome 20
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT- 007)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 29 | 96
EL.U/mL | 573.2 [509.6 to 644.8] | 116.7 [80.9 to 168.3] | 157.5 [128.7 to 192.8]

22. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD) [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 20
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT- 007)
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 264 | 19 | 75
EL.U/mL | 372.4 [329.6 to 420.9] | 144.9 [86.3 to 243.2] | 161.4 [128.4 to 203]

23. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD) [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 20
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 208 | 14 | 54 | 98
EL.U/mL
  Anti-PD antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-PD antibodies, PRE |  |  |  | 106 [91.1 to 123.4]
  Anti-PD antibodies, D7 | 2106 [1806.7 to 2454.9] | 718.2 [442.5 to 1165.7] | 680.7 [522.9 to 886.2] | 382.9 [320.7 to 457.2]
  Anti-PD antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-PD antibodies, M3 |  |  |  | 708.6 [604.6 to 830.4]

24. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any occurrence of symptom regardless of intensity grade. Any Redness or any Swelling symptom = any symptom greater than (>) 0 millimeter (mm). Grade 3 pain = maximum intensity of local injection defined as subject crying when limb was moved/spontaneously painful. Grade 3 redness/swelling= maximum intensity of local injection >30 mm. Follow-up period was of 4 days (Days 0-3) after Synflorix vaccination in Year 4 Persistence and Immunological Memory 111347 Study, thus one period of 4 days for primed subjects and 2 periods of 4 days for unprimed subjects.
Time Frame: Within 4 days (Days 0-3) period(s) after Synflorix vaccination in Year 4 Persistence and Immunological Memory 111347 Study
Population: The analyses were performed on the Total Vaccinated Cohort (TVC) which included all vaccinated subjects. The TVC for analysis of safety included all primed subjects with additional vaccine dose administration documented and all unprimed subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 264 | 20 | 64 | 100
Participants
  Pain, Any | 157 | 9 | 34 | 54
  Redness, Any | 90 | 5 | 14 | 21
  Swelling, Any | 67 | 4 | 15 | 20
  Pain, Grade 3 | 7 | 1 | 5 | 3
  Redness, Grade 3 (> 30 mm) | 7 | 0 | 0 | 1
  Swelling, Grade 3 (> 30 mm) | 5 | 0 | 1 | 2

25. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite and fever (any fever defined as temperature by axillary measurement of 37.5°C and above). Grade 3 drowsiness was defined as drowsiness that prevented normal activity; Grade 3 irritability was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as subject not eating at all. Grade 3 fever was defined as axillary temperature >39.5°C. Related AE was defined as any AE assessed by investigators to be causally related to administration of the study vaccine. Follow-up period was of 4 days (Days 0-3) after Synflorix vaccination in Year 4 Persistence and Immunological Memory 111347 Study, thus one period of 4 days for primed subjects and 2 periods of 4 days for unprimed subjects.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 263 | 20 | 64 | 100
Participants
  Drowsiness, Any | 49 | 2 | 12 | 12
  Drowsiness, Grade 3 | 1 | 0 | 0 | 0
  Drowsiness, Related | 48 | 2 | 11 | 11
  Irritability, Any | 35 | 4 | 6 | 8
  Irritability, Related | 35 | 4 | 6 | 8
  Irritability, Grade 3 | 0 | 0 | 0 | 0
  Loss of appetite, Any | 30 | 3 | 6 | 13
  Loss of appetite, Grade 3 | 1 | 0 | 1 | 0
  Loss of appetite, Related | 30 | 3 | 5 | 11
  Fever, Any | 13 | 0 | 2 | 5
  Fever, >39,5°C | 0 | 0 | 0 | 0
  Fever, Related | 13 | 0 | 1 | 5

26. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination. Follow-up period was of 31 days (Days 0-30) after Synflorix vaccination in Year 4 Persistence and Immunological Memory 111347 Study, thus one period of 31 days for primed subjects and 2 periods of 31 days for unprimed subjects.
Time Frame: Within 31 days (Day 0-30) after Synflorix vaccination in Year 4 Persistence and Immunological Memory 111347 Study
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 264 | 20 | 65 | 100
Participants | 25 | 0 | 3 | 6

27. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to Study Procedures [Follow-up Period: Year 1 (111345 Sub-study)]
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above. "Any" was defined an incidence of a SAE regardless of intensity/severity.
Time Frame: During Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007) i.e. for each primed subject: from the time the subject was enrolled in the 111345 study until he/she completed the same study (approximatively 12 months)
Population: The analysis was performed on the primed subjects who were enrolled in the applicable 111345 Year 1 Follow-Up Study.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 391 | 31 | 102
Participants | 1 | 0 | 0

28. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to Study Procedures [(Follow-up Period: Year 2 (111346 Sub-study) Until Year 4 (111347 Sub-study)]
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above. "Any" is defined an incidence of a SAE regardless of intensity/severity.
Time Frame: From Year (Y) 2 to Y4 FU visit (post booster vaccination administered in 10PN-PD-DIT-007) i.e. for each subject(S): when S was enrolled in 111346 study until S completed the same study visit or the 111347 study visit (range of 1 to 3 years for each S))
Population: The analysis was performed on the Total enrolled cohort which included all primed subjects from Y2 follow-up sub-study 111346 and from Y4 long-term follow-up sub-study 111347 for antibody persistence for whom data concerning antibody persistence were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 370 | 31 | 96
Participants | 0 | 0 | 0

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) [Follow-up Period: Vaccination Period in Year 4 (111347 Sub-study)]
Description: as for outcome 28
Time Frame: For primed groups: from Months 48-49 (additional vaccination period); for unprimed group: from Day 0 up to Month 3 (catch-up vaccination period)
Population: The analyses were performed on the Total Vaccinated Cohort (TVC) which included all vaccinated subjects in study 111347. The TVC for analysis of safety included all primed subjects with additional vaccine dose administration documented and all unprimed subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 264 | 20 | 65 | 100
Participants | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Serotypes [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The seropositivity cut-off for the assay was 8.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 359 | 27 | 94
Participants
  Anti-1 OPA, Y1: number analyzed (Participants) | 354 | 27 | 92
  Anti-1 OPA, Y1 | 188 | 2 | 26
  Anti-4 OPA, Y1: number analyzed (Participants) | 340 | 26 | 86
  Anti-4 OPA, Y1 | 201 | 21 | 65
  Anti-5 OPA, Y1: number analyzed (Participants) | 335 | 27 | 89
  Anti-5 OPA, Y1 | 241 | 2 | 46
  Anti-6B OPA, Y1: number analyzed (Participants) | 354 | 25 | 88
  Anti-6B OPA, Y1 | 164 | 23 | 44
  Anti-7F OPA, Y1: number analyzed (Participants) | 346 | 25 | 89
  Anti-7F OPA, Y1 | 343 | 20 | 85
  Anti-9V OPA, Y1: number analyzed (Participants) | 352 | 26 | 94
  Anti-9V OPA, Y1 | 351 | 26 | 90
  Anti-14 OPA, Y1: number analyzed (Participants) | 343 | 25 | 91
  Anti-14 OPA, Y1 | 336 | 25 | 89
  Anti-18C OPA, Y1: number analyzed (Participants) | 319 | 24 | 84
  Anti-18C OPA, Y1 | 173 | 10 | 25
  Anti-19F OPA, Y1: number analyzed (Participants) | 359 | 27 | 93
  Anti-19F OPA, Y1 | 306 | 19 | 83
  Anti-23F OPA, Y1: number analyzed (Participants) | 336 | 27 | 93
  Anti-23F OPA, Y1 | 301 | 26 | 82

31. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Serotypes [Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: as for outcome 30
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The According-To-Protocol (ATP) cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 354 | 27 | 92
Participants
  Anti-1 OPA, Y2 | 92 | 0 | 15
  Anti-4 OPA, Y2: number analyzed (Participants) | 335 | 27 | 84
  Anti-4 OPA, Y2 | 146 | 12 | 48
  Anti-5 OPA, Y2: number analyzed (Participants) | 351 | 27 | 91
  Anti-5 OPA, Y2 | 169 | 2 | 31
  Anti-6B OPA, Y2: number analyzed (Participants) | 342 | 27 | 88
  Anti-6B OPA, Y2 | 241 | 24 | 67
  Anti-7F OPA Titers, Y2: number analyzed (Participants) | 350 | 27 | 91
  Anti-7F OPA Titers, Y2 | 350 | 26 | 90
  Anti-9V OPA, Y2: number analyzed (Participants) | 349 | 27 | 92
  Anti-9V OPA, Y2 | 347 | 27 | 87
  Anti-14 OPA, Y2: number analyzed (Participants) | 341 | 25 | 90
  Anti-14 OPA, Y2 | 333 | 24 | 85
  Anti-18C OPA, Y2: number analyzed (Participants) | 325 | 27 | 83
  Anti-18C OPA, Y2 | 165 | 11 | 29
  Anti-19F OPA, Y2: number analyzed (Participants) | 349 | 27 | 92
  Anti-19F OPA, Y2 | 279 | 21 | 78
  Anti-23F OPA, Y2: number analyzed (Participants) | 342 | 26 | 91
  Anti-23F OPA, Y2 | 285 | 25 | 72

32. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Serotypes [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 30
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: The According-To-Protocol (ATP) cohort for persistence included all primed subjects from the Total enrolled cohort who had not received a vaccine or product forbidden in the protocol and for whom assay results available for the antibodies against at least one vaccine antigen component for the blood sampling taken at Year 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 250 | 16 | 72
Participants
  Anti-1 OPA, Y4 | 55 | 1 | 17
  Anti-4 OPA, Y4: number analyzed (Participants) | 232 | 16 | 63
  Anti-4 OPA, Y4 | 107 | 8 | 33
  Anti-5 OPA, Y4: number analyzed (Participants) | 243 | 15 | 68
  Anti-5 OPA, Y4 | 80 | 2 | 11
  Anti-6B OPA, Y4: number analyzed (Participants) | 250 | 16 | 68
  Anti-6B OPA, Y4 | 223 | 15 | 62
  Anti-7F OPA, Y4: number analyzed (Participants) | 249 | 15 | 71
  Anti-7F OPA, Y4 | 248 | 15 | 71
  Anti-9V OPA, Y4: number analyzed (Participants) | 250 | 15 | 70
  Anti-9V OPA, Y4 | 242 | 14 | 68
  Anti-14 OPA, Y4: number analyzed (Participants) | 250 | 15 | 71
  Anti-14 OPA, Y4 | 247 | 14 | 70
  Anti-18C OPA, Y4: number analyzed (Participants) | 226 | 16 | 63
  Anti-18C OPA, Y4 | 121 | 8 | 27
  Anti-19F OPA, Y4: number analyzed (Participants) | 247 | 16 | 69
  Anti-19F OPA, Y4 | 211 | 14 | 62
  Anti-23F OPA, Y4: number analyzed (Participants) | 239 | 15 | 65
  Anti-23F OPA, Y4 | 209 | 15 | 55

33. Secondary Outcome: Number of Seropositive Subjects for Opsophagocytic Activity Against Pneumococcal Serotypes [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Analysis was performed with Unprimed group included. The seropositivity cut-off for the assay was 8.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 201 | 13 | 51 | 96
Participants
  Anti-1 OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-1 OPA, PRE |  |  |  | 8
  Anti-1 OPA, D7: number analyzed (Participants) | 197 | 13 | 50 | 92
  Anti-1 OPA, D7 | 193 | 13 | 48 | 90
  Anti-1 OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-1 OPA, M3 |  |  |  | 87
  Anti-4 OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 81
  Anti-4 OPA, PRE |  |  |  | 17
  Anti-4 OPA, D7: number analyzed (Participants) | 196 | 13 | 51 | 93
  Anti-4 OPA, D7 | 194 | 13 | 50 | 93
  Anti-4 OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-4 OPA, M3 |  |  |  | 94
  Anti-5 OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-5 OPA, PRE |  |  |  | 8
  Anti-5 OPA, D7: number analyzed (Participants) | 193 | 13 | 48 | 91
  Anti-5 OPA, D7 | 186 | 13 | 47 | 87
  Anti-5 OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-5 OPA, M3 |  |  |  | 89
  Anti-6B OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 79
  Anti-6B OPA, PRE |  |  |  | 35
  Anti-6B OPA, D7: number analyzed (Participants) | 198 | 13 | 50 | 93
  Anti-6B OPA, D7 | 196 | 13 | 48 | 84
  Anti-6B OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-6B OPA, M3 |  |  |  | 94
  Anti-7F OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 74
  Anti-7F OPA, PRE |  |  |  | 67
  Anti-7F OPA, D7: number analyzed (Participants) | 199 | 13 | 50 | 93
  Anti-7F OPA, D7 | 199 | 13 | 50 | 93
  Anti-7F OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 93
  Anti-7F OPA, M3 |  |  |  | 93
  Anti-9V OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 87
  Anti-9V OPA, PRE |  |  |  | 75
  Anti-9V OPA, D7: number analyzed (Participants) | 201 | 13 | 51 | 93
  Anti-9V OPA, D7 | 201 | 13 | 51 | 93
  Anti-9V OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 94
  Anti-9V OPA, M3 |  |  |  | 94
  Anti-14 OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 83
  Anti-14 OPA, PRE |  |  |  | 81
  Anti-14 OPA, D7: number analyzed (Participants) | 197 | 13 | 51 | 94
  Anti-14 OPA, D7 | 197 | 13 | 51 | 94
  Anti-14 OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-14 OPA, M3 |  |  |  | 95
  Anti-18C OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 89
  Anti-18C OPA, PRE |  |  |  | 7
  Anti-18C OPA, D7: number analyzed (Participants) | 194 | 13 | 50 | 92
  Anti-18C OPA, D7 | 190 | 13 | 48 | 88
  Anti-18C OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-18C OPA, M3 |  |  |  | 92
  Anti-19F OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-19F OPA, PRE |  |  |  | 30
  Anti-19F OPA, D7: number analyzed (Participants) | 196 | 13 | 50 | 93
  Anti-19F OPA, D7 | 194 | 13 | 50 | 91
  Anti-19F OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 93
  Anti-19F OPA, M3 |  |  |  | 93
  Anti-23F OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 83
  Anti-23F OPA, PRE |  |  |  | 47
  Anti-23F OPA, D7: number analyzed (Participants) | 199 | 13 | 50 | 96
  Anti-23F OPA, D7 | 197 | 13 | 49 | 95
  Anti-23F OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-23F OPA, M3 |  |  |  | 95

34. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 6A and 19A. The results for the immune responses were measured by 22F-inhibition ELISA. The seropositivity cut-off for the assay was 0.05 μg/mL.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 390 | 31 | 102
Participants
  Anti-6A antibodies, Y1 | 376 | 31 | 97
  Anti-19A antibodies, Y1 | 366 | 29 | 93

35. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 6A and 19A. The immune responses were measured by 22F-inhibation ELISA. The seropositivity cut-off for the assay was 0.05 μg/mL.
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 30 | 96
Participants
  Anti-6A antibodies, Y2 | 330 | 30 | 86
  Anti-19A antibodies, Y2 | 319 | 25 | 83

36. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 6A and 19A. The immune responses were measured by 22F-inhibition ELISA. The seropositivity cut-off for the assay was 0.05 μg/mL.
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 263 | 19 | 75
Participants
  Anti-6A antibodies, Y4: number analyzed (Participants) | 263 | 19 | 74
  Anti-6A antibodies, Y4 | 256 | 18 | 72
  Anti-19A antibodies, Y4 | 260 | 18 | 74

37. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 36
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 208 | 14 | 54 | 98
Participants
  Anti-6A antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-6A antibodies, PRE |  |  |  | 76
  Anti-6A antibodies, D7 | 208 | 14 | 54 | 92
  Anti-6A antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-6A antibodies, M3 |  |  |  | 97
  Anti-19A antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-19A antibodies, PRE |  |  |  | 88
  Anti-19A antibodies, D7 | 208 | 14 | 54 | 97
  Anti-19A antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-19A antibodies, M3 |  |  |  | 98

38. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 6A and 19A. The immune responses were mesured by Opsonophagocytic activity (OPA). The seropositivity cut-off for the assay was 8.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 352 | 26 | 93
Participants
  Anti-6A OPA, Y1: number analyzed (Participants) | 323 | 25 | 75
  Anti-6A OPA, Y1 | 196 | 24 | 45
  Anti-19A OPA, Y1 | 45 | 3 | 10

39. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 2 (111346 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. Pneumococcal serotypes assessed were 6A and 19A. The immune responses were measured by Opsonophagocytic activity (OPA). The seropositivity cut-off for the assay was 8.
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 351 | 27 | 91
Participants
  Anti-6A OPA, Y2: number analyzed (Participants) | 314 | 25 | 82
  Anti-6A OPA, Y2 | 235 | 21 | 62
  Anti-19A OPA, Y2 | 115 | 8 | 29

40. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 39
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 246 | 15 | 68
Participants
  Anti-6A OPA Titers, Y4: number analyzed (Participants) | 231 | 14 | 66
  Anti-6A OPA Titers, Y4 | 194 | 12 | 51
  Anti-19A OPA Titers, Y4 | 135 | 7 | 34

41. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes 6A and 19A [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 39
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 194 | 13 | 49 | 92
Participants
  Anti-6A OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 82
  Anti-6A OPA, PRE |  |  |  | 57
  Anti-6A OPA, D7: number analyzed (Participants) | 189 | 12 | 49 | 92
  Anti-6A OPA, D7 | 185 | 12 | 46 | 88
  Anti-6A OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 91
  Anti-6A OPA, M3 |  |  |  | 87
  Anti-19A OPA, PRE: number analyzed (Participants) | 0 | 0 | 0 | 92
  Anti-19A OPA, PRE |  |  |  | 25
  Anti-19A OPA, D7: number analyzed (Participants) | 194 | 13 | 48 | 90
  Anti-19A OPA, D7 | 173 | 11 | 36 | 81
  Anti-19A OPA, M3: number analyzed (Participants) | 0 | 0 | 0 | 91
  Anti-19A OPA, M3 |  |  |  | 87

42. Secondary Outcome: Number of Seropositive Subjects for Anti-protein D (Anti-PD) [Follow-up Period: Persistence Analysis in Year 1 (111345 Sub-study)]
Description: A seropositive subject was a subject whose anti-PD antibody concentration was greater than or equal to (≥) the cut-off value. The seropositivity cut-off for the assay was 100 EL.U/ML.
Time Frame: At Year 1 (Y1) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 390 | 30 | 102
Participants | 373 | 11 | 71

43. Secondary Outcome: Number of Seropositive Subjects for Anti Protein D (Anti-PD) [Follow-up Period: Persistence Analysis in Year 2 (111345 Sub-study)]
Description: as for outcome 42
Time Frame: At Year 2 (Y2) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 368 | 29 | 96
Participants | 340 | 15 | 65

44. Secondary Outcome: Number of Seropositive Subjects for Anti-protein D (Anti-PD) [Follow-up Period: Persistence Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 42
Time Frame: At Year 4 (Y4) (post booster vaccination administered in study 10PN-PD-DIT-007)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix
Number analyzed (Participants) | 261 | 19 | 74
Participants | 241 | 12 | 54

45. Secondary Outcome: Number of Seropositive Subjects for Anti-protein D (Anti-PD) [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the cut-off value. The seropositivity cut-off for the assay was 100 EL.U/ML.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 208 | 14 | 54 | 98
Participants
  Anti-PD antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 95
  Anti-PD antibodies, PRE |  |  |  | 54
  Anti-PD antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 96
  Anti-PD antibodies, D7 | 207 | 14 | 54 | 92
  Anti-PD antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-PD antibodies, M3 |  |  |  | 98

46. Secondary Outcome: Number of Seropositive Subjects for Anti-vaccine Pneumococcal Serotypes Antibodies [Follow-up Period: Immunogenicity Analysis in Year 4 (111347 Sub-study)]
Description: as for outcome 1
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
Number analyzed (Participants) | 208 | 14 | 54 | 98
Participants
  Anti-1 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-1 antibodies, PRE |  |  |  | 69
  Anti-1 antibodies, D7 | 207 | 14 | 54 | 97
  Anti-1 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-1 antibodies, M3 |  |  |  | 98
  Anti-4 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-4 antibodies, PRE |  |  |  | 29
  Anti-4 antibodies, D7 | 208 | 14 | 54 | 98
  Anti-4 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-4 antibodies, M3 |  |  |  | 98
  Anti-5 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-5 antibodies, PRE |  |  |  | 72
  Anti-5 antibodies, D7 | 207 | 14 | 54 | 98
  Anti-5 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-5 antibodies, M3 |  |  |  | 98
  Anti-6B antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-6B antibodies, PRE |  |  |  | 77
  Anti-6B antibodies, D7: number analyzed (Participants) | 208 | 14 | 54 | 97
  Anti-6B antibodies, D7 | 207 | 14 | 54 | 94
  Anti-6B antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-6B antibodies, M3 |  |  |  | 98
  Anti-7F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-7F antibodies, PRE |  |  |  | 64
  Anti-7F antibodies, D7 | 208 | 14 | 54 | 98
  Anti-7F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-7F antibodies, M3 |  |  |  | 98
  Anti-9V antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-9V antibodies, PRE |  |  |  | 67
  Anti-9V antibodies, D7 | 208 | 14 | 54 | 94
  Anti-9V antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-9V antibodies, M3 |  |  |  | 98
  Anti-14 antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-14 antibodies, PRE |  |  |  | 90
  Anti-14 antibodies, D7 | 208 | 14 | 54 | 97
  Anti-14 antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-14 antibodies, M3 |  |  |  | 98
  Anti-18C antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-18C antibodies, PRE |  |  |  | 52
  Anti-18C antibodies, D7 | 207 | 14 | 54 | 97
  Anti-18C antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-18C antibodies, M3 |  |  |  | 98
  Anti-19F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 96
  Anti-19F antibodies, PRE |  |  |  | 75
  Anti-19F antibodies, D7 | 208 | 14 | 54 | 97
  Anti-19F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-19F antibodies, M3 |  |  |  | 98
  Anti-23F antibodies, PRE: number analyzed (Participants) | 0 | 0 | 0 | 97
  Anti-23F antibodies, PRE |  |  |  | 54
  Anti-23F antibodies, D7 | 208 | 14 | 54 | 90
  Anti-23F antibodies, M3: number analyzed (Participants) | 0 | 0 | 0 | 98
  Anti-23F antibodies, M3 |  |  |  | 98

ADVERSE EVENTS:
Time Frame: Solicited and Unsolicited AEs were collected within 4 days and 31 days post-Synflorix vaccination, respectively, for subjects participating to Year 4 follow-up period. SAEs related to study procedure were collected at Year 1 in sub-study 111345 and from Year 2 up to Year 4 follow-up period in sub-studies 111346-111347 for primed subjects. Any SAEs were collected during the vaccination period in the111347 study (i.e. from Month 48-49 for primed subjects and from Month 0-3 for unprimed subjects).
Arm/Group | Synflorix + Infanrix + Havrix and/or Varilrix Group | Prevenar + Infanrix + Havrix and/or Varilrix Group | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix | Unprimed Group
All-Cause Mortality (participants affected / at risk) | 0/391 | 0/31 | 0/102 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/391 | 0/31 | 0/102 | 0/100
Other Adverse Events (participants affected / at risk) | 188/264 | 12/20 | 39/65 | 65/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix + Infanrix + Havrix and/or Varilrix Group (N=391) | Prevenar + Infanrix + Havrix and/or Varilrix Group (N=31) | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix (N=102) | Unprimed Group (N=100)
Broncopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix + Infanrix + Havrix and/or Varilrix Group (N=264) | Prevenar + Infanrix + Havrix and/or Varilrix Group (N=20) | Prevenar + Synflorix + Infanrix + Havrix and/or Varilrix (N=65) | Unprimed Group (N=100)
Pain (General disorders) | 157 | 9 | 34/64 | 54
Redness (General disorders) | 90 | 5 | 14/64 | 21
Swelling (General disorders) | 67 | 4 | 15/64 | 20
Drowsiness (General disorders) | 49/263 | 2 | 12/64 | 12
Irritability (General disorders) | 35/263 | 4 | 6/64 | 8
Loss of appetite (General disorders) | 30/263 | 3 | 6/64 | 13
Fever (Axillary temperature ≥ 37.5°C) (General disorders) | 13/263 | 0 | 2/64 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.